CLINICAL TRIAL: NCT01170793
Title: Medication Overuse Headaches: the Impact of Educative Telephone Coaching Administered by Nurses Prior to the Medical Appointment in a Tertiary Consultation Center: a Comparative Randomized Trial
Brief Title: Medicine Abuse Headache
Acronym: CAM-ET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2009/16
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Migraine
Keywords: education, quality of life
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (No Intervention): no educative telephone coaching (ETC)
- 1 (Experimental): with educative telephone coaching (ETC)
  Interventions: Behavioral: educative telephone coaching (ETC)

INTERVENTIONS:
Behavioral: educative telephone coaching (ETC) — a 30 to 45 minutes phone call, by appointment, by the nurse
  Arms: 1

SUMMARY:
In patients with MOH, we will evaluate the impact of educative telephone coaching on the number of days with headache over the month preceding the appointment. The educative coaching will be administered by a nurse, during a single phone call and prior to the medical visit

DETAILED DESCRIPTION:
In tertiary centers, it is not unusual for patients to wait for 6 months for a medical appointment. This clinical trial is monocentric, open, randomised. In the first arm, the patients will receive educative telephone coaching at Month 2 by the nurses, over the phone. In the second arm, the patients will not receive any educative telephone coaching before the appointment with the neurologist.

All patients will complete "Quality of life" questionnaires at Month 1 and Months 6, complete a migraine agenda during the length of the study and have a medical appointment around Month 6.

The primary outcome will be the efficacy of such educative telephone coaching, administered before the medical appointment in the Chronic Pain Center, in Bordeaux. It will be measured by the number of days with headache over the month preceding the appointment.

ELIGIBILITY:
Inclusion Criteria:

* Adults, male or female, > 18 years old
* Patients with a presumptive medication overuse headache diagnostic (>15 days/month with migraines, > 10 days/month intake of crisis treatment)
* Persons calling the Chronic Pain Center in Bordeaux and asking for a medical appointment
* Informed and written consent, dated and signed by the patient and the investigator prior to any study related procedure

Exclusion Criteria:

* Patients with a differential diagnostic (other primitive headaches and secondary headaches)
* Persons non affiliated to a social security system
* Persons who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of educative telephone coaching administered by the center's nurses prior to the medical on-site visit. | within 6 months

SECONDARY OUTCOMES:
To evaluate the efficacy of educative telephone coaching (ETC) on the frequency of headaches and on the number of days with crisis treatment intake. | within 6 months
To evaluate the efficacy of ETC on the patients quality of life and their handicap (emotional, professional and familial data) | within 6 months
To evaluate the patient's satisfaction toward ETC | within 6 months
To evaluate the patient's knowledge concerning migraine, medication overuse headache and their treatment after ETC | within 6 months
To estimate the cost/benefits ratio of ETC and its impact on medical costs ahead of the medical appointment. | within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève Chene, MD PhD, Study Chair — University Hospital, Bordeaux; Virginie Dousset, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Centre Douleur Chronique - Groupe Hospitalier Pellegrin - Bât USN Tastet Girard, Bordeaux, France